CLINICAL TRIAL: NCT02533700
Title: CEOP/IVE/GDP Compared With CEOP as the First-line Therapy for Newly Diagnosed Adult Patients With Peripheral T-cell Lymphoma (PTCL)
Brief Title: CEOP/IVE/GDP Compared With CEOP as the First-line Therapy for Newly Diagnosed Adult Patients With PTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Hematology Department, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WXin
Record Dates: First submitted 2015-07-18; First posted 2015-08-27 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Peripheral T-Cell Lymphoma, Not Otherwise Specified; Angioimmunoblastic T Cell Lymphoma; ALK-negative Anaplastic Large Cell Lymphoma; Enteropathy Associated T Cell Lymphoma; Subcutaneous Panniculitis Like T Cell Lymphoma; Hepatosplenic T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Subcutaneous panniculitis-like T-cell lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CEOP/IVE/GDP chemotherapy regimen (Experimental): 2 cycles of CEOP(cyclophosphamide,vincristine, epirubucin and prednisone),2 cycles of IVE(ifosfamide, epirubucin, etoposide)and 2 cycles of GDP(gemcitabine, cis-platinum, and dexamethasone)
  Interventions: Drug: CEOP/IVE/GDP chemotherapy regimen
- CEOP chemotherapy regimen for 6 cycles (Active Comparator): 6 cycles of CEOP regimen(cyclophosphamide,vincristin,epirubucin and prednisone)
  Interventions: Drug: CEOP chemotherapy regimen for 6 cycles

INTERVENTIONS:
Drug: CEOP/IVE/GDP chemotherapy regimen — CEOP:
  Cyclophosphamide 750mg/m2, ivgtt D1 Epirubucin 70mg/m2,ivgtt D1 Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5
  IVE:
  Ifosfamide 2000mg/m2,ivgtt D1-D3 Epirubucin 70mg/m2, ivgtt D1 Etoposide 100mg/m2, ivgtt D1-D3
  GDP:
  Gemcitabine 1g/m2,ivgtt D1,D8 Cis-platinum 25mg/m2, ivgtt D1-D3 Dexamethasone 40mg, ivgtt D1-D4
  Arms: CEOP/IVE/GDP chemotherapy regimen
Drug: CEOP chemotherapy regimen for 6 cycles — CEOP:
  Cyclophosphamide 750mg/m2, ivgtt D1 Epirubucin 70mg/m2,ivgtt D1 Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5 every 21 days for total 6 courses
  Arms: CEOP chemotherapy regimen for 6 cycles

SUMMARY:
Peripheral T-cell Lymphoma (PTCL) is a heterogenic malignancy with poor outcome. Five-year PFS and OS for these patients received classic CHOP regimen (cyclophosphamide, vincristin, doxorubicin and prednisone) is less than 30%.High dose intensive chemotherapy doesn't demonstrate better response. At present, there is no standardized treatment protocol for this kind of lymphoma. So, clinical trials are encouraged by NCCN for those patients.

DETAILED DESCRIPTION:
For the less efficacy of CHOP or CHOP-like regimen, multi-drug combination strategy has been the therapy tendency in PTCL. The novel regimen IVE/MTX (ifosfamide, etoposide，epirubucin/methotrexate)-ASCT(autologous stem-cell transplantation ) was piloted for patients eligible for intensive treatment, followed by auto-stem cell transplantation. Five-years PFS (progression-free survival) and OS (overall survival) were 52% and 60% respectively, significantly improved compared with the historical group treated with anthracycline-based chemotherapy. The encouraged results were extended to the peripheral T cell lymphoma-non specified (PTCL-NOS). Former studies reported that GDP (gemcitabine, cis-platinum, and dexamethasone) compared with CHOP as the therapy strategy for PTCL-NOS (not otherwise specified). The response rate was 78.57% in GDP group and 60.00% in CHOP group respectively. DFS (disease-free survival) was 9.79 and 4.2 months in above two groups. They concluded that GDP is superior with CHOP. The main side-effect of two regimens is hematological toxicity. Furthermore, high-dose combined with ASCT has been the first-line therapy for PTCL. However, only about 30% patients with PTCL have chance to receive ASCT for multiple reasons. So it is urgent to explore new combination-therapy regimen to improve the outcome for patients with PTCL.

The aim of our study is to compare the response and survival rate of CEOP/IVE/GDP (cyclophosphamide, vincristin, epirubucin and prednisone/ ifosfamide, epirubucin, and etoposide/ gemcitabine, cis-platinum, and dexamethasone) with those of CEOP regimen, looking forward to its superiority in efficacy and safety for the newly diagnosed adult patients with PTCL.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically confirmed the following pathology subtype according to WHO 2008 classification: peripheral T Cell Lymphoma, not otherwise specified, angioimmunoblastic T cell lymphoma, ALK-negative anaplastic large cell lymphoma, enteropathy associated T cell lymphoma, subcutaneous panniculitis like T cell lymphoma, and hepatosplenic T-cell lymphoma.
* ≥ 16 years of age.
* Performance status of 2 or less.
* Has no history of malignancy.
* Has radiologically measurable disease.
* Life expectancy ≥6 months.
* Voluntarily sign an informed consent.

Exclusion Criteria:

* Pathology subtype with NK/T cell lymphoma, ALK positive-ALCL.
* Primary central nervous system (CNS) lymphoma.
* Previous systemic chemotherapy or local therapy.
* Has undergone hematopoietic stem-cell transplantation (HSCT).
* Has active infectious disease requiring general antibiotics, anti-fungal or anti-virus therapy.
* Has uncontrollable cardiocerebrovascular, coagulative, autoimmune, or serious infectious disease.
* Echocardiography shows left ventricular ejection fraction (LVEF) ≤ 50%.
* Inadequate renal, hepatic or bone marrow function
* Active liver or biliary disease.
* Has other uncontrollable medical condition that may interfere with their participation in the study.
* Woman in pregnancy or lactation.
* Patient is known to be positive for Human immunodeficiency virus (HIV) infection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete remission （CR） | 6 months

SECONDARY OUTCOMES:
progression-free survival | 2 year since randomization
overall survival | 2 year since randomization
overall response rate | 6 months
adverse events | from randomization to one month after last cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, PhD, Principal Investigator — Shanghai Province Hopsital
Locations (4):
- China (4):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Cai MC, Cheng S, Wang X, Hu JD, Song YP, Huang YH, Yan ZX, Jiang YJ, Fang XS, Zheng XY, Dong LH, Ji MM, Wang L, Xu PP, Zhao WL. CEOP/IVE/GDP alternating regimen compared with CEOP as the first-line therapy for newly diagnosed patients with peripheral T cell lymphoma: results from a phase 2, multicenter, randomized, controlled clinical trial. Genome Med. 2020 Apr 30;12(1):41. doi: 10.1186/s13073-020-00739-0. PMID 32349779